CLINICAL TRIAL: NCT02904876
Title: Evaluation of Early Changes Visible to the Diffusion MRI in Response to Two Years of Treatment With Tysabri in Patients With Multiple Sclerosis
Acronym: TYSADIFF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5815
Record Dates: First submitted 2014-12-08; First posted 2016-09-19 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnetic Resonance Imaging at 6 months (Experimental): 2-year follow-up MRI of patients initiating treatment with Tysabri with anti-JCV antibody positive or negative. Patients enrolled will benefit from diffusion MRI at 6 months, in addition to conventional MRI.
  Interventions: Radiation: Diffusion Magnetic Resonance Imaging at 6 months

INTERVENTIONS:
Radiation: Diffusion Magnetic Resonance Imaging at 6 months — 2-year follow-up MRI of patients initiating treatment with Tysabri with anti-JCV antibody positive or negative. Patients enrolled will benefit from diffusion MRI at 6 months, in addition to conventional MRI.

SUMMARY:
Through this phase IV study, multicenter prospective exploratory, uncontrolled, the investigators propose to identify MRI predictive factors of treatment response, using diffusion MRI sequences, in addition to conventional sequences.

The primary objective is to study the links between changes on MRI diffusion and response to treatment with Tysabri to 2 years.

The secondary objective is to compare the evolution of diffusion MRI data with the volumetric MRI data.

ELIGIBILITY:
Inclusion Criteria:

* Major Patient
* Patient with relapsing remitting multiple sclerosis and eligible for treatment with Tysabri
* Patient affiliated to a social security scheme
* Patient who signed informed consent
* Patient who have been informed of the results of the prior medical examination

Exclusion Criteria:

* Patient not currently eligible for treatment with Tysabri
* Contraindication to MRI scanning
* Unability to provide informed consent (subject in an emergency situation, difficulties in understanding , ...)
* Patient under judicial protection
* Patient under guardianship or curatorship
* Pregnancy (women of childbearing age in the absence of effective contraception)
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Comparaison of diffusion Magnetic Resonance Imaging before and after the initiation of treatment with Tysabri using fractional anisotropy (FA). | 24 months

SECONDARY OUTCOMES:
Comparison of different Magnetic Resonance Imaging criteria before and after treatment | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme DE SEZE, Principal Investigator — Service de Neurologie HUS hautepierre
Locations (1):
- Service de Neurologie Hôpital de Hautepierre, Strasbourg, Alsace, France